CLINICAL TRIAL: NCT00847119
Title: ESTUDIO FASE II DE BEVACIZUMAB EN COMBINACIÓN CON CAPECITABINA Y RADIOTERAPIA COMO TRATAMIENTO PREOPERATORIO EN PACIENTES CON CÁNCER RECTAL LOCALMENTE AVANZADO RESECABLE
Brief Title: Xeloda and Bevacizumab to Treat Rectal Cancer
Acronym: xeberecto
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML 20006. XEBERECTO/ICO/005; EudraCT number:2007-000456-13
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Rectal Cancer
Keywords: rectum; adenocarcinoma; neoadjuvant; bevacizumab; capecitabine; radiotherapy; locally; advanced; resectable; resectable locally advanced adenocarcinoma of the rectum; xeberecto
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma | interventions — Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab & capecitabine & radiotheraphy (Experimental): Bevacizumab 4 cycles each 15 days, the first 10 mg/kg and the rest of cycles with 5 mg/kg.
  Radiotherapy 45 Gy starting on Bevacizumab 2nd cycle during 5 weeks, 1.8 Gy per day, 5 days at week.
  Capecitabine 900 mg/m2 two times a day concomitant during radiotherapy period.
  Interventions: Biological: Bevacizumab; Drug: capecitabine (Xeloda); Radiation: Rectal Radiotherapy

INTERVENTIONS:
Biological: Bevacizumab — Bevacizumab 4 cycles each 15 days, the first 10 mg/kg and the rest of cycles with 5 mg/kg.
Drug: capecitabine (Xeloda) — Capecitabine 900 mg/m2 two times a day concomitant during radiotherapy period
Radiation: Rectal Radiotherapy — Radiotherapy in rectum 45 Gy starting on Bevacizumab 2nd cycle during 5 weeks, 1.8 Gy per day, 5 days at week.

SUMMARY:
The project objective is to evaluate the efficacy of the neoadjuvant treatment with bevacizumab, capecitabine and radiotherapy, in patients with rectal adenocarcinoma resectable locally advanced (stage T3 or T4), with or without presence of ganglionar metastases and without distant metastases.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has given written informed consent prior to any study related procedure
2. Male and female aged 18 to 75 years
3. ECOG performance status 0 or 1
4. Histologically confirmed diagnostic of adenocarcinoma of the rectum < 15 cm from anal verge
5. Clinical stage of T3, T4 with/without regional lymph node metastases, without metastatic disease
6. Disease evaluable by imaging techniques
7. No tumour haemorrhage in the week prior to start of study treatment
8. External derivation in symptomatic occlusive tumours
9. Not prior cancer treatment
10. Adequate bone marrow, hepatic and renal function, defined as:

    1. White blood cells ≥ 4 x 109 /l
    2. Absolute neutrophil count ≥ 1.5 x 109 /l
    3. Platelets ≥ 100 x 109 /l
    4. Haemoglobin ≥10 g/dl
    5. Bilirubin < 1.25 x upper limit of normal
    6. Aspartate transaminase and alanine transaminase < 2.5 x upper limit of normal
    7. Serum creatinine ≤ 106 µmol/l
11. Less than 10% weight loss

Exclusion Criteria:

1. Rectal cancer no amenable to resection
2. Any other malignancy which has been active or treated within the past 5 years , with the exception of in situ carcinoma of the cervix and non-melanoma skin lesions adequately treated
3. Pregnant or breast-feeding women
4. Women oh childbearing potential unless effective methods of contraception are used
5. No prior or concurrent significant medical conditions, including any of the following:

   * Cerebrovascular disease (including transient ischemic attack and stroke) within the past year
   * Cardiovascular disease, including the following:
   * Myocardial infarction within the past year
   * Uncontrolled hypertension while receiving chronic medication
   * Unstable angina
   * New York Heart Association class II-IV congestive heart failure
   * Serious cardiac arrhythmia requiring medication
6. Major trauma within the past 28 days
7. Serious nonhealing wound, ulcer, or bone fracture
8. Evidence of bleeding diathesis or coagulopathy
9. No lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication
10. No evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug
11. No known dihydropyrimidine dehydrogenase deficiency
12. Major surgery in the 4 weeks prior to the start of study treatment
13. No concurrent chronic, daily treatment with aspirin (> 325 mg/day)
14. More than 10 days since prior use of full-dose oral or parenteral anticoagulants for therapeutic purposes
15. No participation in another clinical trial with any investigational drug within 30 days prior to randomization or during study participation
16. No other medical history or condition that, in the opinion of the investigator, would preclude study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response rate. % patients with pathologic complete response (absence of tumoral cells in the resected piece) | Surgery date

SECONDARY OUTCOMES:
Overall clinical response | Surgery date
To determine the downstaging caused by treatment | Surgery date
relapse free survival | Time of radiological evidence of relapse.
Quantify the local control grade: R0 resections in surgery | Surgery date
Local relapse and distant relapse rates | Relapse date
To determine the security profile of this neoadjuvant treatment (radio- chemotherapy) | From date of register to surgery date
Surgery complication rate | During surgery admission.
To determine the angiogenic profile changes in tumour. | 15 days, 6 weeks and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Salazar, Phd, Principal Investigator — Institut Català d'Oncologia; Margarita Garcia, MD, Study Chair — Institut Català d'Oncologia
Locations (1):
- Institut Català d'Oncologia-L'Hospitalet, L'Hospitalet Del Llobregat, Barcelona, Spain

REFERENCES:
- [Result] Garcia M, Martinez-Villacampa M, Santos C, Navarro V, Teule A, Losa F, Pisa A, Cambray M, Soler G, Lema L, Kreisler E, Figueras A, Juan XS, Vinals F, Biondo S, Salazar R. Phase II study of preoperative bevacizumab, capecitabine and radiotherapy for resectable locally-advanced rectal cancer. BMC Cancer. 2015 Feb 26;15:59. doi: 10.1186/s12885-015-1052-0. PMID 25886275